CLINICAL TRIAL: NCT05885555
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Ianalumab (VAY736) in Patients With Primary Immune Thrombocytopenia (ITP) Previously Treated With at Least a Corticosteroid and a Thrombopoietin Receptor Agonist (TPO-RA)
Brief Title: A Study of Ianalumab (VAY736) in Patients With Primary Immune Thrombocytopenia (ITP) Previously Treated With at Least Two Lines of Therapies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAY736Q12201; 2022-503041-21-00 (Other: EU CTIS)
Expanded Access: NCT07244289 (Available)
Record Dates: First submitted 2023-05-15; First posted 2023-06-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: Primary immune thrombocytopenia (ITP); ianalumab; VAY736; B-cell depletion; B-cell Activating Factor Receptor (BAFF-R) blockade
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — ianalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): All eligible participants will receive ianalumab at the same dose.
  Interventions: Biological: Ianalumab

INTERVENTIONS:
Biological: Ianalumab — Intravenous infusion, prepared from concentrate solution
  Other Names: VAY736

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy, safety and tolerability of ianalumab in adult patients with primary ITP previously treated with at least one corticosteroid and one TPO-RA.

DETAILED DESCRIPTION:
This is a phase 2, open-label, single-arm study to evaluate the efficacy, safety and tolerability of ianalumab in participants with primary ITP (platelet count <30 G/L at screening) previously treated with at least a corticosteroid and a TPO-RA.

The study consists of the screening period, the primary endpoint assessment period, the follow-up period. The screening period will last for up to 14 days prior to the first dose of ianalumab. All eligible participants will be treated with the same dose of ianalumab and will complete the primary endpoint assessment period. After completion of the primary endpoint assessment period, all participants will continue in safety monitoring and those with a platelet count ≥30 G/L in absence of a new line of ITP therapy and rescue therapy will also continue in efficacy monitoring. The trial includes an option to offer a second course of ianalumab treatment to participants who achieved confirmed response during the initial course of ianalumab and later lost response to explore the benefit of the second course of treatment. The study will end once all participants have completed 24 months of safety follow-up since their last dose of ianalumab (including the optional second course of ianalumab treatment),or discontinued the study earlier.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to participation in the study.
* Male or female participants aged 18 years and older on the day of signing informed consent.
* Confirmed diagnosis of primary ITP.

  * Prior treatment with at least a corticosteroid (±IVIG) and a TPO-RA:
  * Prior additional therapies are allowed; the corticosteroid or the TPO-RA do not need to be the last treatment.
  * Prior response to IVIG/anti-D or a corticosteroid (platelet count ≥50 G/L) that was not maintained.
* At last ITP treatment, loss of response, insufficient response, no response or intolerance.
* Platelet count <30 G/L and assessed as needing treatment (per physician's discretion) at screening. If concomitant ITP medication is clinically indicated, the platelet assessment showing a value <30 G/L must be performed after at least 14 days on a stable dose of a corticosteroid or/and a TPO-RA (less than 10% variation from current dose) and continue stable thereafter.

Key exclusion criteria:

* Diagnosis of secondary thrombocytopenia.
* Platelet or whole blood transfusion, plasmapheresis, or use of any other rescue medications within 14 days before first ianalumab infusion.
* Participants with the following conditions at screening:

  * Neutrophils <1000/mm3.
  * Immunoglobulin G (IgG) <5 g/L
* Treatment with a B-cell depleting therapy (e.g., rituximab) or anti-B-cell Activating Factor of the TNF Family (BAFF) (e.g., belimumab) within 12 weeks prior to the first administration of ianalumab.
* Immunosuppressant drugs other than corticosteroids within 5 times the elimination half-life of the drug or 14 days before first ianalumab infusion, whichever is longer.
* Prior splenectomy.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2029-03-19 (Estimated)

PRIMARY OUTCOMES:
Confirmed response | Between Week 1 Day 1 and Week 25 Day 1
  Confirmed response is defined as a platelet count of equal or above 50 G/L at two (or more) consecutive assessments at least 7 days apart, in the absence of:
  * Rescue treatment for ≥4 weeks prior to the assessment of the platelet count, and
  * New immune thrombocytopenia (ITP) treatment before reaching a confirmed response.

SECONDARY OUTCOMES:
Time to confirmed response | From Week 1 Day 1 to Week 25 Day 1
  Time from the first administration of ianalumab to the first assessment in the first sequence of two (or more) platelet assessments meeting the criteria of a confirmed response as defined by the primary endpoint.
Duration of confirmed response | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Time from the first assessment in the first sequence of two (or more) platelet assessments meeting the criteria of a confirmed response to loss of response; with loss of response defined as the first of the following events:
  * platelet count <30 G/L,
  * start of any rescue or new ITP treatment,
  * death (whatever the cause).
Complete Response rate at each timepoint | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Percentage of participants with a platelet count of at least 100 G/L in the absence of rescue treatment/new ITP treatment.
Response rate at each timepoint | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Percentage of participants with a platelet count of at least 50 G/L in the absence of rescue treatment/new ITP treatment.
Stable response at 6 months | At 6 months
  Percentage of participants with at least 75% of platelet counts collected at month 6 (between study days 121 and 183) equal to or above 50 G/L in the absence of rescue treatment/new ITP treatment.
Stable response at 1 year | At 1 year
  Percentage of participants with at least 66% of platelet counts collected at year 1 (between study days 296 and 379) equal to or above 50 G/L in the absence of rescue treatment/new ITP treatment.
Bleeding events according to the Modified World Health Organization (WHO) bleeding scale | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Number of participants reporting bleeding events for each grade of the World Health Organization (WHO) bleeding scale at each time point. Severity is graded from 0 to 4, with 0 = no bleeding and 4 = severe hemodynamic instability/central nervous system (CNS) bleeding/fatal.
Percentage of participants with bleeding events according to the Modified World Health Organization (WHO) bleeding scale | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Percentage of participants reporting bleeding events for each grade of the WHO bleeding scale at each time point. Severity is graded from 0 to 4, with 0 = no bleeding and 4 = severe hemodynamic instability/central nervous system (CNS) bleeding/fatal.
Number of participants who received rescue treatment | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Number of participants who required rescue treatment
Percentage of participants who received rescue treatment | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Percentage of participants who required rescue treatment
Change from baseline in the frequency of CD19+ B-cell counts | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Post-baseline frequency of CD19+ B-cell counts compared to baseline
Change from baseline in the absolute number of CD19+ B-cell counts | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Post-baseline absolute number of CD19+ B-cell counts compared to baseline
Time to first occurrence of B-cell recovery defined as ≥80% of baseline ≥50 cells/µL | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Time to B-cell recovery defined as ≥80% of baseline or ≥50 cells/µL
Change from baseline in immunoglobulins | From Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Post-baseline immunoglobulin levels (change in titers of Total Ig, IgG, IgM, IgA) compared to baseline
Incidence of anti-ianalumab antibodies in serum (ADA assay) over time | Up to 20 weeks after last dose of ianalumab
  Anti-drug antibodies (ADA) will be evaluated in samples collected from all participants to assess the immunogenicity of ianalumab
Titer of anti-ianalumab antibodies in serum (ADA assay) over time | Up to 20 weeks after last dose of ianalumab
  Anti-drug antibodies (ADA) will be evaluated in samples collected from all participants to assess the immunogenicity of ianalumab
Ianalumab serum concentrations over time | First dose (pre-dose, 2, 168, 336, 504, 672 hours post-dose); Subsequent doses (pre-dose and 2 hours post-dose); Last dose (pre-dose, 2 336, 672, 1344, 2016, 3360 hours post-dose)
  Ianalumab concentration in serum over time, including end of infusion and concentration at trough.
Ianalumab serum PK: AUC concentrations over time | First dose (pre-dose, 2, 168, 336, 504, 672 hours post-dose); Subsequent doses (pre-dose and 2 hours post-dose); Last dose (pre-dose, 2 336, 672, 1344, 2016, 3360 hours post-dose)
  Ianalumab concentration in serum over time, including end of infusion and concentration at trough.
Ianalumab serum PK parameters: Cmax | First dose (pre-dose, 2, 168, 336, 504, 672 hours post-dose); Subsequent doses (pre-dose and 2 hours post-dose); Last dose (pre-dose, 2 336, 672, 1344, 2016, 3360 hours post-dose)
  Maximum (peak) observed plasma, blood, serum or other body fluid drug concentration
Ianalumab serum PK parameters: Tmax | First dose (pre-dose, 2, 168, 336, 504, 672 hours post-dose); Subsequent doses (pre-dose and 2 hours post-dose); Last dose (pre-dose, 2 336, 672, 1344, 2016, 3360 hours post-dose)
  Time to reach maximum (peak) observed plasma, blood, serum or other body fluid drug concentration
Confirmed response (CR) in the second course | Second course Week 1 Day1 to second course Week 25 Day1
  Confirmed response is defined as a platelet count of equal or above 50 G/L at two (or more) consecutive assessments at least 7 days apart, in the absence of:
  * Rescue treatment for ≥4 weeks prior to the assessment of the platelet count, and
  * New ITP treatment before reaching a confirmed response.
Time to confirmed response in the second course | Second course Week 1 Day 1 to second course Week 25 Day 1
  two (or more) platelet assessments meeting the criteria of a confirmed response.
Duration of confirmed response in the second course | Second course Week 1 Day 1 to second course Week 25 Day 1
  Time from the first assessment, in the second course of two (or more) platelet assessments meeting the criteria of a confirmed response to loss of response; with loss of response defined as the first of the following events:
  * platelet count <30 G/L,
  * start of any rescue or new ITP treatment,
  * death (whatever the cause).
Response in the second course | Second course Week 1 Day 1 to second course Week 25 Day 1
  Percentage of participants with a platelet count of at least 50 G/L in the absence of rescue treatment/new ITP treatment.
Complete Response in the second course | Second course Week 1 Day 1 to second course Week 25 Day 1
  Percentage of participants with a platelet count of at least 100 G/L in the absence of rescue treatment/new ITP treatment.
Bleeding events in the second course according to the Modified World Health Organization (WHO) bleeding scale | Second course Week 1 Day 1 to second course Week 25 Day 1
  Number of participants reporting bleeding events for each grade of the World Health Organization (WHO) bleeding scale at each time point. Severity is graded from 0 to 4, with 0 = no bleeding and 4 = severe hemodynamic instability/central nervous system (CNS) bleeding/fatal.
Percentage of participants with bleeding events in the retreatment/second courseaccording to the Modified World Health Organization (WHO) bleeding scale | Second course Week 1 Day 1 to second course Week 25 Day 1
  Percentage of participants reporting bleeding events for each grade of the WHO bleeding scale at each time point. Severity is graded from 0 to 4, with 0 = no bleeding and 4 = severe hemodynamic instability/central nervous system (CNS) bleeding/fatal.
Number of Participants who received rescue treatment after second course | Second course Week 1 Day 1 to second course Week 25 Day 1
  Number of participants who required rescue treatment
Percentage of participants who received rescue treatment after receiving second course | Second course Week 1 Day 1 to second course Week 25 Day 1
  Percentage of participants who required rescue treatment
Titer of anti-ianalumab antibodies in serum (ADA assay) over time for second course | Second course Week 1 Day 1 until 20 weeks after last dose of ianalumab
  Anti-drug antibodies (ADA) will be evaluated in samples collected from all participants to assess the immunogenicity of ianalumab
Change from start of second course in immunoglobulins | From second course Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Post-baseline immunoglobulin levels (change in titers of Total Ig, IgG, IgM, IgA) compared to retreatment baseline
Change from start of second course in the absolute number of CD19+ B-cell counts | From second course Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Post-baseline absolute number of CD19+ B-cell counts compared to baseline
Change from start of second course to end of study in the absolute number of CD19+ B-cell counts | From second course Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Post-baseline absolute number of CD19+ B-cell counts compared to baseline
Time to first occurrence of B-cell recovery defined as ≥80% of baseline ≥50 cells/µL | From second course Week 1 Day 1 to end of study (until all participants have completed 24 months of safety follow-up since their last dose of ianalumab or discontinued the study earlier)
  Time to B-cell recovery defined as ≥80% of baseline or ≥50 cells/µL
Ianalumab serum concentrations over time in the second course | First dose (pre-dose, 2, 168, 336, 504, 672 hours post-dose); Subsequent doses (pre-dose and 2 hours post-dose); Last dose (pre-dose, 2 336, 672, 1344, 2016, 3360 hours post-dose) in the second course
  Ianalumab concentration in serum over time, including end of infusion and concentration at trough.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Med Center, Boston, Massachusetts
- Novartis Investigative Site, CABA, Argentina
- Australia (2):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Melbourne, Victoria
- China (3):
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Jinan
- Novartis Investigative Site, Toulouse, France
- Germany (3):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Giessen
- Novartis Investigative Site, Torino, TO, Italy
- Novartis Investigative Site, Johor Bahru, Malaysia
- Novartis Investigative Site, Katowice, Poland
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Aydin, Efeler
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Edirne, Merkez
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
- United Kingdom (2):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com